CLINICAL TRIAL: NCT07115108
Title: Effectiveness of High-Energy Density Enteral Nutrition for Enhancing Physical Growth and Cognitive Brain Development in Infants With Congenital Heart Disease: A Randomized Controlled Study
Brief Title: Effectiveness of High-Energy Density Enteral Nutrition for Enhancing Physical Growth and Cognitive Brain Development in Infants With Congenital Heart Disease
Acronym: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNF; 2024YFC707605 (Other Grant/Funding Number: National Health Commission of the People's Republic of China)
Record Dates: First submitted 2025-07-30; First posted 2025-08-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Congenital Heart Disease; Enteral Nutrition; Pediatrics
Keywords: Congenital heart disease; Enteral nutrition; Pediatrics
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High energy density enteral nutrition (Experimental): High-energy-density enteral nutrition (100 cal/100 ml) will be administered to infants following surgery for congenital heart disease. The target feeding volume will be determined based on the infant's body weight (80-100 ml/kg), with the volume per feeding and frequency appropriately adjusted. Weight measurements and neurological assessments will be conducted at admission, prior to discharge, and at 1-, 3-, and 6-month intervals post-discharge. The safety of the intervention will be closely monitored throughout the study period.
  Interventions: Dietary Supplement: High energy density enteral nutrition
- General energy density enteral nutrition (Active Comparator): General energy density enteral nutrition (60-88cal/100 ml) will be administered to infants following surgery for congenital heart disease. The target feeding volume will be determined based on the infant's body weight (80-100 ml/kg), with the volume per feeding and frequency appropriately adjusted. Weight measurements and neurological assessments will be conducted at admission, prior to discharge, and at 1-, 3-, and 6-month intervals post-discharge. The safety of the intervention will be closely monitored throughout the study period.
  Interventions: Dietary Supplement: General energy density enteral nutrition

INTERVENTIONS:
Dietary Supplement: High energy density enteral nutrition — High-energy-density enteral nutrition (100 cal/100 ml) will be administered to infants following surgery for congenital heart disease. The target feeding volume will be determined based on the infant's body weight (80-100 ml/kg), with the volume per feeding and frequency appropriately adjusted.
  Other Names: High energy density EN
  Arms: High energy density enteral nutrition
Dietary Supplement: General energy density enteral nutrition — General energy density enteral nutrition (60-88 cal/100 ml) will be administered to infants following surgery for congenital heart disease. The target feeding volume will be determined based on the infant's body weight (80-100 ml/kg), with the volume per feeding and frequency appropriately adjusted.
  Other Names: General energy density EN
  Arms: General energy density enteral nutrition

SUMMARY:
The purpose of this study is to compare the effect of high and ordinary energy density enteral nutrition for improving physical growth and brain cognitive development in infants with congenital heart disease after operation, as well as evaluate the safety of interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital heart disease through symptoms, physical signs, imaging, and ultrasound examinations.
* Age 0-6 months
* Children with nutritional risks (defined by STRONGkids: Nutritional risk screening tool for children )
* Artificial or mixed feeding
* Open heart surgery under cardiopulmonary bypass
* The guardians of the children voluntarily participate in this study and sign a written informed consent form before the surgery.

Exclusion Criteria:

* Diagnosed with major non cardiac diseases leading to nutritional intake disorders, such as congenital gastrointestinal malformations, preoperative diagnosis of gastroesophageal reflux, genetic diseases related to growth restriction, and various syndromes with chromosomal abnormalities (trisomy 21 syndrome, trisomy 18 syndrome)
* Abnormal immune system function due to congenital or acquired factors, unable to effectively resist pathogens or eliminate abnormal cells, which can be divided into primary and secondary immunodeficiencies.
* Any pre - operative history of neurological diseases (e.g., encephalitis, epilepsy).
* Secondary or primary gastrointestinal infection symptoms such as abdominal distension and diarrhea after surgery.
* Estimated stay time in the postoperative intensive care unit ≤ 2 days

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight-for-age z score (WAZ) | 6th month after discharge
  WAZ is calculated according to the Chinese child growth curve and cut-offs .It is a statistical index used to assess the nutritional status of children. The physical examination will be conducted by a nurse, and the data will be recorded to one decimal place.

SECONDARY OUTCOMES:
Weight-for-age z score (WAZ) | Before discharge, 1st month, 3rd month after discharge
  WAZ is calculated according to the Chinese child growth curve and cut-offs .It is a statistical index used to assess the nutritional status of children. The physical examination will be conducted by a nurse, and the data will be recorded to one decimal place.
Cognitive development | Before discharge, 1st month, 3rd month, 6th month after discharge
  The Griffiths mental development scales (GMDs) will be used to repeatedly measure the indicators .The Griffiths scales typically yield a Developmental Quotient (DQ) with an average range of 85-115. The higher the scores, the more advanced development relative to age norms in assessed domains (e.g., motor, language, or cognition).
Incidence of subjects with Gastrointestinal mucosal barrier function injury | Before discharge, 1 month, 3 months, 6 months after discharge
  Primarily defined by elevation in fecal calprotectin and Inflammatory cytokines level.The reference range for calprotectin is 0-5 μg/g，inflammatory cytokines is ≤20pg/ml.Exceeding this range will be considered as abnormal gastrointestinal mucosal barrier function.
Albumin level | Before discharge, 1 month, 3 months, 6 months after discharge
  Albumin is a rich protein in the blood, which mainly reflects the nutritional status.The reference range for albumin is 39-54g/L.If it is not within this range, it will be judged as abnormal.
Blood lipid levels | Before discharge, 1 month, 3 months, 6 months after discharge
  Blood lipid test is to measure the content of lipids in blood.Blood lipids include total cholesterol(0-5.18mmol/L) and triglycerides(0-1.7mmol/L).If it exceeds the range, it will be considered as abnormal.
Energy intake (cal/d) | During hospitalization, before discharge, 1 month, 3 months, 6 months after discharge
  Calculate the caloric intake for enteral feeding according to the Schofeld formula recommended by the European Society for Pediatric and Neonatal Intensive Care (ESPNIC)
Enteral Nutrition intake (ml/d) | During hospitalization, before discharge, 1 month, 3 months, 6 months after discharge
  Based on the child's weight and the fluid balance in the previous 24 hours, the total fluid intake for the day is calculated. After subtracting the amount of intravenous drug solution, the amount of enteral nutrition formula is obtained. According to the child's gastrointestinal function, the principle of gradual progress is adopted to rationally allocate the single feeding volume and feeding frequency.
Incidence of malabsorption | During hospitalization, before discharge, 1 month, 3 months, 6 months after discharge
  Incidence of malabsorption (as defined by any of the following criteria): abnormal fecal lactose content; abnormal fecal fat content.The diagnosis will be confirmed by fecal examination.
Incidence of feeding intolerance | During hospitalization, before discharge, 1 month, 3 months, 6 months after discharge
  Any of the following condition: 1. Frequent vomiting (≥ 3 times/d); 2.Abdominal distension; 3. Milk volume did not increase or decreased>3 d; 4. Gastric retention (retention>1/3 of the previous feeding); 5. Unplanned discontinuation of feeding ≥ 2 times; 6. Diarrhea (stool frequency>6 times/d)
Incidence of necrotizing enterocolitis（NEC） | Before discharge, 1 month, 3 months, 6 months after discharge
  NEC diagnosed in stage II and III will be recorded.
Other surgical indications | At the day of discharge, an average of 3 week after surgery
  Mechanical ventilation time (days), postoperative CCU hospitalization duration (days), total hospitalization duration (days), hospitalization costs (Yuan), and the incidence of poor wound healing will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region